CLINICAL TRIAL: NCT01828047
Title: Correlation Between Sublingual Microcirculation and Postoperative Ileus Symptoms in Patients Undergoing Colorectal Surgery - a Pilot Study
Brief Title: Sublingual Microcirculation and Postoperative Ileus
Status: Completed | Type: Observational
Sponsor: Gabriele Baldini, MD, MSc, Assistant Professor (Other)
Responsible Party: Sponsor-Investigator, Gabriele Baldini, MD, MSc, Assistant Professor, Assitant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Other Study IDs: 12-214-SDR
Record Dates: First submitted 2012-10-31; First posted 2013-04-10 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Colorectal Cancer; Inflammatory Bowel Diseases; Gastrointestinal Dysfunction
MeSH Terms: conditions — Colorectal Neoplasms; Inflammatory Bowel Diseases | interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective colorectal surgeries: Patients undergoing elective colorectal procedures with an Enhanced Recovery Program. Orthogonal polarization spectral (OPS) imaging will be used to measure sublingual microcirculation
  Interventions: Device: orthogonal polarization spectral (OPS) imaging

INTERVENTIONS:
Device: orthogonal polarization spectral (OPS) imaging — orthogonal polarization spectral (OPS) imaging allows noninvasive observation of human microcirculation in all accessible tissue surfaces

SUMMARY:
The aim of this pilot study is to establish if a correlation between sub-lingual microcirculation measured by Orthogonal polarization spectral (OPS) imaging and symptoms of postoperative ileus exist in patients undergoing elective colorectal surgery.

DETAILED DESCRIPTION:
AIM OF THE STUDY This observational study will assess whether perioperative microcirculatory changes can be correlated with symptoms associated with primary POI.

PRIMARY RESEARCH QUESTION Is there a correlation between peri-operative microcirculatory flow measurements and the incidence of symptomatic primary POI?

SECONDARY RESEARCH QUESTIONS

1. Is there a correlation between peri-operative microcirculatory flow measurements and the duration of symptomatic primary POI?
2. If any correlation is observed, which anatomic location (sublingual mucosa vs bowel serosa) yields microcirculatory flow measurements that are more strongly associated with the incidence and/or duration of symptomatic primary POI?
3. Can either intraoperative sublingual mucosa or intraoperative bowel serosa microcirculatory flow measurements predict symptoms of primary POI? Are these two anatomic locations equivalent in their ability to predict this complication?

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 yo undergoing elective laparoscopic colorectal surgery with an Enhanced Recovery Program (ERP) at the Montreal General Hospital

Exclusion Criteria:

* Any patient who refuses enrolment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective colorectal surgery with an Enhanced Recovery Program (ERP)
Sampling Method: Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2013-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Postoperative ileus symptoms; microvascular flow index (MFI) | Participants will be followed for the duration of hospital stay, an expected average of 3 days
  Patients will be considered having POI symptoms if at least one symptom, for each of the following criteria, will be reported:
  i. Vomiting (+/- nausea) OR abdominal distension AND ii. Absence of passing gas/stool OR not tolerating oral diet.
  Microvascular flow index (MFI) score: this score is based on determination of the predominant type of flow observed. Flow is characterized as absent (0), intermittent (1), sluggish (2), or normal (3).

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Baldini, MD, MSc, Principal Investigator — McGill University
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Kehlet H. Multimodal approach to postoperative recovery. Curr Opin Crit Care. 2009 Aug;15(4):355-8. doi: 10.1097/MCC.0b013e32832fbbe7. PMID 19617822
- [Background] Kehlet H. Postoperative ileus--an update on preventive techniques. Nat Clin Pract Gastroenterol Hepatol. 2008 Oct;5(10):552-8. doi: 10.1038/ncpgasthep1230. Epub 2008 Aug 12. PMID 18695704
- [Background] Hasibeder W. Gastrointestinal microcirculation: still a mystery? Br J Anaesth. 2010 Oct;105(4):393-6. doi: 10.1093/bja/aeq236. No abstract available. PMID 20837720
- [Background] Bezemer R, Bartels SA, Bakker J, Ince C. Clinical review: Clinical imaging of the sublingual microcirculation in the critically ill--where do we stand? Crit Care. 2012 Jun 19;16(3):224. doi: 10.1186/cc11236. PMID 22713365
- [Background] Jhanji S, Lee C, Watson D, Hinds C, Pearse RM. Microvascular flow and tissue oxygenation after major abdominal surgery: association with post-operative complications. Intensive Care Med. 2009 Apr;35(4):671-7. doi: 10.1007/s00134-008-1325-z. Epub 2008 Oct 21. PMID 18936911
- [Background] Cassina T, Santambrogio L. Microcirculation after cardiopulmonary bypass: a glance at the mesenteric mucosa. Minerva Anestesiol. 2012 Mar;78(3):288-90. No abstract available. PMID 22357370
- [Background] De Backer D, Dubois MJ, Schmartz D, Koch M, Ducart A, Barvais L, Vincent JL. Microcirculatory alterations in cardiac surgery: effects of cardiopulmonary bypass and anesthesia. Ann Thorac Surg. 2009 Nov;88(5):1396-403. doi: 10.1016/j.athoracsur.2009.07.002. PMID 19853081
- [Background] Wongyingsinn M, Baldini G, Charlebois P, Liberman S, Stein B, Carli F. Intravenous lidocaine versus thoracic epidural analgesia: a randomized controlled trial in patients undergoing laparoscopic colorectal surgery using an enhanced recovery program. Reg Anesth Pain Med. 2011 May-Jun;36(3):241-8. doi: 10.1097/AAP.0b013e31820d4362. PMID 21519309
- [Background] Carli F, Charlebois P, Baldini G, Cachero O, Stein B. An integrated multidisciplinary approach to implementation of a fast-track program for laparoscopic colorectal surgery. Can J Anaesth. 2009 Nov;56(11):837-42. doi: 10.1007/s12630-009-9159-x. Epub 2009 Jul 29. PMID 19639371
- [Background] Puhl G, Schaser KD, Vollmar B, Menger MD, Settmacher U. Noninvasive in vivo analysis of the human hepatic microcirculation using orthogonal polorization spectral imaging. Transplantation. 2003 Mar 27;75(6):756-61. doi: 10.1097/01.TP.0000056634.18191.1A. PMID 12660497
- [Background] Rauchfuss F, Scheuerlein H, Ludewig S, Uberruck T, Heise M, Zanow J, Settmacher U. In vivo assessment of the hepatic microcirculation after mesenterico-portal bypass (REX-shunt) using orthogonal polarization spectral imaging. Liver Int. 2010 Oct;30(9):1339-45. doi: 10.1111/j.1478-3231.2010.02311.x. PMID 20666991
- [Background] De Backer D, Hollenberg S, Boerma C, Goedhart P, Buchele G, Ospina-Tascon G, Dobbe I, Ince C. How to evaluate the microcirculation: report of a round table conference. Crit Care. 2007;11(5):R101. doi: 10.1186/cc6118. PMID 17845716
- [Background] Vignali A, Gianotti L, Braga M, Radaelli G, Malvezzi L, Di Carlo V. Altered microperfusion at the rectal stump is predictive for rectal anastomotic leak. Dis Colon Rectum. 2000 Jan;43(1):76-82. doi: 10.1007/BF02237248. PMID 10813128
- [Background] Trzeciak S, Rivers EP. Clinical manifestations of disordered microcirculatory perfusion in severe sepsis. Crit Care. 2005;9 Suppl 4(Suppl 4):S20-6. doi: 10.1186/cc3744. Epub 2005 Aug 25. PMID 16168070
- [Background] Lewis SJ, Egger M, Sylvester PA, Thomas S. Early enteral feeding versus "nil by mouth" after gastrointestinal surgery: systematic review and meta-analysis of controlled trials. BMJ. 2001 Oct 6;323(7316):773-6. doi: 10.1136/bmj.323.7316.773. PMID 11588077
- [Background] Moore FA, Feliciano DV, Andrassy RJ, McArdle AH, Booth FV, Morgenstein-Wagner TB, Kellum JM Jr, Welling RE, Moore EE. Early enteral feeding, compared with parenteral, reduces postoperative septic complications. The results of a meta-analysis. Ann Surg. 1992 Aug;216(2):172-83. doi: 10.1097/00000658-199208000-00008. PMID 1386982
- [Background] Giglio MT, Marucci M, Testini M, Brienza N. Goal-directed haemodynamic therapy and gastrointestinal complications in major surgery: a meta-analysis of randomized controlled trials. Br J Anaesth. 2009 Nov;103(5):637-46. doi: 10.1093/bja/aep279. PMID 19837807